CLINICAL TRIAL: NCT05444036
Title: Caudal Ketamine-bupivacaine More Effective Than Bupivacaine-saline in Pediatric Surgical Procedures Below the Umbilicus
Brief Title: Caudal Ketamine-bupivacaine More Effective Than Bupivacaine-saline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIRVANA 2
Record Dates: First submitted 2022-06-21; First posted 2022-07-05 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-06

CONDITIONS: Surgery; Pediatric Surgery
Keywords: Caudal bupivacaine; ketamine; anaesthesia; paediatric surgeries
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: comparing caudal block by bupivacaine with and without ketamine in paediatric patients undergoing surgery below the umbilicus with regard to analgesic, anaesthetic, and sedative properties.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamin-bupivacaine Group (Experimental): in this method,30 patients which received 0.5 mg/kg of preservative free ketamine (i.e. 0.05ml/kg of 10mg/ml ketamine diluted up to 1ml in normal saline) plus1ml/kg of 0.25 % bupivacaine caudally, after induction of general anaesthesia
  Interventions: Drug: Ketamine
- bupivacaine-saline Group (Experimental): 30 patients received 1ml/kg of 0.25 % bupivacaine plus 1ml of normal saline caudally of just after induction of general anaesthesia, just after induction of general anaesthesia
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — compare caudal ketamine-bupivacaine against caudal bupivacaine-saline in paediatric Measuring pain in patients undergoing surgery below the umbilicus with regard to analgesic, anaesthetic, and sedative properties

SUMMARY:
Because pain is difficult to measure in children, post-operative pain is frequently undertreated in this age range. Pain treatment is required in children due to the high emotional component of pain. Pain is a multidimensional, subjective, perceptual event having a variety of qualities such as intensity, quality, time course, and effects that are perceived differently by each person. Because the operational definition of pain necessitates self-report, pain experienced by children and babies is frequently overlooked, if not ignored.

When general anesthesia is paired with regional procedures, children of all ages are exposed to less intravenous and inhalational anesthetics and analgesics, leaving them nearly free of nausea, vomiting, itching, or unneeded drowsiness. Being completely awake and able to drink soon after surgery, as well as having no issues breathing even after lengthy surgery, are significant benefits that children and parents value.

DETAILED DESCRIPTION:
Caudal block provides the potential benefit of extending the length and effectiveness of the block by combining additional medications with the local anaesthetic agent. Morphine, clonidine, ketamine, and midazolam were among the drugs used.

Although peripheral nerve blocks and caudal anesthesia are relatively safe, extreme attention is required to minimize adverse consequences. Pediatric anesthesiologists must have adequate training to ensure patient safety. A well-trained pediatric anesthesiologist will try to avoid unsafe regional anesthetic application methods and will always be prepared to manage dangerous side effects (overdoses, intravenous administration induced seizures, tip displacement of epidural catheters or centrally located abscesses).

Ketamine is a non-competitive N-methyl D-aspartate NMDA receptor antagonist that is thought to prevent or reverse central sensitization and, as a result, lessen postoperative pain. It also has a peripheral analgesic effect.

Ketamine infiltration has been demonstrated to provide pain alleviation in children having adenotonsillectomy for up to 24 hours following surgery with no adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1- All children whom were diagnosed with herniotomy, orchidopexy, or urethroplasty.

Exclusion Criteria:

1. Drugs used allergy or sensitivity,
2. contraindications to caudal injection, such as infection at the injection site,
3. bleeding disorders
4. caudal vertebral abnormalities

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Post-operative Pain | 24-hour analgesic after surgery
  Assessment of the pain post-operatively in Pediatric patients with pain score as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain, measured in millimetres from the left end bar to the mark placed by the kid on the 10 cm line anchored by happy faces (no pain) to sad faces (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana Elshalakany, Professor, Principal Investigator — Department of Anesthesia and I.C.U. faculty of Medicine October six university, Egypt
Locations (1):
- October 6 University Hospital, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided